CLINICAL TRIAL: NCT01766739
Title: Phase I Study of Intra-pleural Administration of GL-ONC1, a Genetically Modified Vaccinia Virus, in Patients With Malignant Pleural Effusion: Primary, Metastases and Mesothelioma
Brief Title: Intra-pleural Administration of GL-ONC1, a Genetically Modified Vaccinia Virus, in Patients With Malignant Pleural Effusion: Primary, Metastases and Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genelux Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-169
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
Keywords: GL-ONC1; pleural effusion; 12-169
MeSH Terms: conditions — Lung Neoplasms; Pleural Effusion

ARMS (1):
- GL-ONC1 (Experimental): This is an open-label, dose-escalating, non-randomized, single-center Phase I therapeutic study of GL-ONC1 originally administered intrapleurally as a single dose and now escalating to three consecutive daily doses in patients with a diagnosis (histologically or cytologically documented) of malignant pleural effusions.
  Interventions: Biological: GL-ONC1

INTERVENTIONS:
Biological: GL-ONC1 — Patients will be enrolled in groups of three and individually assessed for safety and dose limiting toxicity (DLT).

SUMMARY:
The purpose of this study is to test the safety of the GL-ONC1 vaccinia virus at different dose levels. The investigators want to find out what effects, good and/or bad, it has on the patient and the malignant pleural effusion. A malignant pleural effusion is a build up of fluid in the chest cavity cause by the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically documented, malignant pleural effusions (primary non-small-cell lung carcinoma, mesothelioma, and other histologies), who have free pleural space (partial or total) that permits the intrapleural drug instillation. This includes cytologically negative pleural effusion in conjunction with histologically proven malignancy involving the pleura.
* Age must be ≥ 18 years.
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedures must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0) Grade ≤ 1.
* Any surgery, where general anesthesia was administered, must have occurred at least 14 days prior to study enrollment.
* Chemotherapy, radiotherapy or immunotherapy must have stopped more than 7 days prior to receiving study drug; however, small field palliative radiotherapy, TKI therapies and hormonal therapies are allowed.
* Patients with stage IV malignancy (non-mesothelioma) must have had a brain scan (MRI or CT with contrast) showing no evidence of disease progression within 8 weeks of study enrollment.
* ECOG Zubrod ≤ 2.
* Required baseline laboratory data include:
* Absolute neutrophil count (ANC) ≥ 1.5 × 109 [SI units 10^9/L],
* Platelets ≥ 100 ×10^9 [SI units 10^9/L],
* Hemoglobin ≥ 9.0 g/dL [SI units gm/L],
* Serum creatinine ≤ 1.5 × upper limit of normal (ULN),
* Bilirubin ≤ 1.5 × ULN,
* AST/ALT ≤ 2.5 × ULN (≤ 5 × ULN in the presence of liver metastases)
* Negative pregnancy test for females of childbearing potential.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Patients with fever or any active systemic infections, including known HIV, hepatitis B or C.
* Patients on immunosuppressive therapy or with immune system disorders, including autoimmune diseases.
* Concurrent steroid use of more than an equivalent of 20 mg/day prednisone (or equivalent).
* Prior splenectomy.
* Previous organ transplant.
* Patients with clinically significant dermatological disorders, e.g., eczema or psoriasis, as judged by the principal investigator, or any unhealed skin wounds or ulcers.
* Clinically significant cardiac disease (New York Heart Association, Class III or IV).
* Dementia or altered mental status that would prohibit informed consent.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality, that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results and, in the judgment of the principal investigator, would make the patient inappropriate for this study.
* Known allergy to ovalbumin or other egg products.
* Prior gene therapy treatments or prior therapy with cytolytic virus of any type.
* Concurrent therapy with any other investigational anticancer agent.
* Concurrent antiviral agent active against vaccinia virus (e.g. cidofovir, vaccinia immunoglobulin) during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 2 years
  MTD is to provide a dosing recommendation for subsequent Phase II studies. Three patients will be enrolled in each cohort at the dose levels shown in the table below in order to determine the Maximum Tolerated Dose (MTD). At the beginning of a new dose level, only one patient will be treated. The first patient in each cohort must be treated and complete 14 days of post-treatment evaluation prior to the treatment of the remaining two patients in that cohort.

SECONDARY OUTCOMES:
safety | 2 years
  The safety, tolerability and feasibility of GL-ONC1 will be assessed by the evaluation of the type, frequency, and severity of adverse events (AEs), changes in clinical laboratory tests (hematological and chemistry), immunogenicity and physical examination. All AEs and laboratory toxicities will be graded on the CTCAE (version 4).
detection of virus in body fluids | days 2, 3, 4, & 5. pretreatment
  Patients will undergo serial sampling of blood, sputum, urine samples and pleural drainage for evaluation of viral particles by VPA immediately before treatment, and on days 2, 3, 4 and 5 pretreatment.
evaluation of viral appearance in tumor | 2-9 days after intrapleural instillation of virus
  Unless medically contraindicated, patients will undergo Video-Assisted Thoracic Surgery (VATS) with pleural biopsies to assess for green fluorescent protein (GFP) viral expression in tumor and surrounding tissues, and if appropriate, to perform pleurodesis at 2-7 days after intrapleural instillation of virus. Random pleural biopsies and GFP-directed biopsies will be performed to allow for assessment of viral presence. Viral plaque assays (VPA) will be performed in tumor biopsies. Immunohistochemical (IHC) and beta-glucuronidase assay staining for GL-ONC1 will be performed on both GFP (-) and (+) areas at videothoracoscopy (if applicable).
Therapeutic efficacy | day 60 post treatment (+/-10 days)
  Therapeutic efficacy will be investigated with CT scans pretreatment and at Day 60 (+/-10) posttreatment. Response by RECIST criteria (and by modified RECIST - for mesothelioma tumors) will be summarized for each dose level using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Rusch, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Chintala NK, Choe JK, McGee E, Bellis R, Saini JK, Banerjee S, Moreira AL, Zauderer MG, Adusumilli PS, Rusch VW. Correlative analysis from a phase I clinical trial of intrapleural administration of oncolytic vaccinia virus (Olvi-vec) in patients with malignant pleural mesothelioma. Front Immunol. 2023 Feb 16;14:1112960. doi: 10.3389/fimmu.2023.1112960. eCollection 2023. PMID 36875061
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/